CLINICAL TRIAL: NCT04656366
Title: Coronary Angiographical Results in Patients With Angina After CABG: Comparison Between No-touch and Conventional Vein Graft
Brief Title: Results of Coronary Angiography Rafter CABG: Comparison Between No-touch and Conventional Vein Graft
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Gabriele Ferrari, Principal Investigator, Region Örebro County
Other Study IDs: OLL-274418
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Bypass Graft Stenosis
Keywords: vein graft; no-touch; angina; coronary angiography; graft patency
MeSH Terms: conditions — Angina Pectoris | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No-touch: Participants that operated at the time of the coronary artery bypass grafting with a "no-touch" venous graft.
  Interventions: Diagnostic Test: Coronary Angiography
- Conventional: Participants that operated at the time of the coronary artery bypass grafting with a "conventional" venous graft.
  Interventions: Diagnostic Test: Coronary Angiography

INTERVENTIONS:
Diagnostic Test: Coronary Angiography — Diagnostic Coronary angiography for patients that presented angina after a previous CABG operation; eventually interventional procedure with PCI (Percutaneous Coronary Intervention)
  Other Names: Previously: coronary artery bypass grafting (CABG)

SUMMARY:
Coronary artery disease is one of the biggest health issue worldwide: It is estimated that cardiovascular diseases cause around 45% of all death in Sweden and in the West World. The treatment, in a large part of the patients, implicates a so called bypass-operation, that consists in to connect new vascular conduits (grafts) beyond the narrowed coronary vessels to improve the blood supply to the heart. One of the graft that is commonly used is the saphenous vein from the leg. The disadvantage of the saphenous vein graft is the predisposition to early obstruction. The international literature shows the following grades of occlusion: 15% in the first year and 40% after 10 years.

At the Cardio-Thoracic Clinic of the University hospital of Örebro has been developed a new method to harvest the saphenous vein together with the surrounding fat-tissue. This technique, called no-touch technique, has the advantage to reduce the damages to the vein during the harvesting, showing a substantially reduced risk for future occlusion (5% after 18 months and 10% after 8,5 years).

2020-05-20 2020-11-16 Project created in: FoU Region Örebro län Resultat av Koronarangiografi hos patienter som tidigare CABG opererats Project number : 274418 Created by: Gabriele Ferrari, 2020-05-20 Last revised by: Gabriele Ferrari, 2020-11-16 Ongoing The aim of the PhD project is to evaluate the results of the no-touch technique in compare to the conventional technique for the venous graft harvesting. The focus of the study is to analyze all the operated patients in our clinic who underwent a post-operative coronary angiography do to angina pectoris (heart pain). One will compare the patency rate, the rate of MACE (major adverse cardiac events) and the quality of life in the two groups (no-touch vs. conventional). This study is the first and the only one in the world that will examine the long-term angiographic results of the no-touch technique in patients that had angina pectoris after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Angina after CABG requiring diagnostic coronary angiography
* CABG operation between 1992 and June 30th 2020
* Coronary angiography between 2006 and June 30th 2020

Exclusion Criteria:

* Coronary angiography within 30 days from the CABG operation date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the subjects that previously were operated with a coronary artery bypass grafting at the Cardiothoracic department of the University hospital of Orebro (from1992 until June 30th 2020) and that underwent a percutaneous coronary intervention in a venous graft between January the 1st, 2006 and June the 30th, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Graft Patency | after the primary CABG (until June the 30th 2020)
  Grade of freedom from stenosis in the saphenous vein graft used during the primary CABG

SECONDARY OUTCOMES:
Rate of MACE | after the primary CABG (until June the 30th 2020)
  major adverse cardiac events

CONTACTS AND LOCATIONS:
Locations (1):
- Kärl-Thoraxkliniken; University Hospital of Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Souza D. A new no-touch preparation technique. Technical notes. Scand J Thorac Cardiovasc Surg. 1996;30(1):41-4. doi: 10.3109/14017439609107239. No abstract available. PMID 8727856
- [Background] Souza DS, Dashwood MR, Tsui JC, Filbey D, Bodin L, Johansson B, Borowiec J. Improved patency in vein grafts harvested with surrounding tissue: results of a randomized study using three harvesting techniques. Ann Thorac Surg. 2002 Apr;73(4):1189-95. doi: 10.1016/s0003-4975(02)03425-2. PMID 11996262
- [Background] Souza DS, Johansson B, Bojo L, Karlsson R, Geijer H, Filbey D, Bodin L, Arbeus M, Dashwood MR. Harvesting the saphenous vein with surrounding tissue for CABG provides long-term graft patency comparable to the left internal thoracic artery: results of a randomized longitudinal trial. J Thorac Cardiovasc Surg. 2006 Aug;132(2):373-8. doi: 10.1016/j.jtcvs.2006.04.002. PMID 16872965
- [Background] Samano N, Geijer H, Bodin L, Arbeus M, Mannion JD, Dashwood M, Souza D. The no-touch saphenous vein graft in elderly coronary bypass patients with multiple comorbidities is a promising conduit to substitute the left internal thoracic artery. J Thorac Cardiovasc Surg. 2017 Aug;154(2):457-466.e3. doi: 10.1016/j.jtcvs.2017.03.048. Epub 2017 Mar 24. PMID 28433355
- [Background] Bourassa MG. Fate of venous grafts: the past, the present and the future. J Am Coll Cardiol. 1991 Apr;17(5):1081-3. doi: 10.1016/0735-1097(91)90835-w. No abstract available. PMID 2007707
- [Background] Hindnavis V, Cho SH, Goldberg S. Saphenous vein graft intervention: a review. J Invasive Cardiol. 2012 Feb;24(2):64-71. PMID 22294536
- [Background] Goldman S, Zadina K, Moritz T, Ovitt T, Sethi G, Copeland JG, Thottapurathu L, Krasnicka B, Ellis N, Anderson RJ, Henderson W; VA Cooperative Study Group #207/297/364. Long-term patency of saphenous vein and left internal mammary artery grafts after coronary artery bypass surgery: results from a Department of Veterans Affairs Cooperative Study. J Am Coll Cardiol. 2004 Dec 7;44(11):2149-56. doi: 10.1016/j.jacc.2004.08.064. PMID 15582312
- [Background] Lee MS, Park SJ, Kandzari DE, Kirtane AJ, Fearon WF, Brilakis ES, Vermeersch P, Kim YH, Waksman R, Mehilli J, Mauri L, Stone GW. Saphenous vein graft intervention. JACC Cardiovasc Interv. 2011 Aug;4(8):831-43. doi: 10.1016/j.jcin.2011.05.014. PMID 21851895
- [Background] Stone GW, Goldberg S, O'Shaughnessy C, Midei M, Siegel RM, Cristea E, Dangas G, Lansky AJ, Mehran R. 5-year follow-up of polytetrafluoroethylene-covered stents compared with bare-metal stents in aortocoronary saphenous vein grafts the randomized BARRICADE (barrier approach to restenosis: restrict intima to curtail adverse events) trial. JACC Cardiovasc Interv. 2011 Mar;4(3):300-9. doi: 10.1016/j.jcin.2010.11.013. PMID 21435608
- [Derived] Ferrari G, Loayza R, Azari A, Geijer H, Cao Y, Carlsson R, Bojo L, Samano N, Souza D. Superior long-term patency of no-touch vein graft compared to conventional vein grafts in over 1500 consecutive patients. J Cardiothorac Surg. 2024 Oct 1;19(1):570. doi: 10.1186/s13019-024-03057-3. PMID 39354611